CLINICAL TRIAL: NCT02096029
Title: Brief, Novel Smoking Cessation in Primary Care: A Comparative Effectiveness Trial
Brief Title: Tobacco Intervention in Primary Care Treatment Opportunities for Providers
Acronym: TipTop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Matthew Carpenter, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00019201; 2R01DA021619 (NIH)
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Smoking; Smoking Cessation
Keywords: smoking; smoking cessation; nicotine replacement therapy; primary care; comparative effectiveness
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Nicotine Replacement Therapy; corticosteroid hormone-induced factor; Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicotine Replacement Therapy (NRT) (Experimental): 2 week supply of 4 mg nicotine lozenge and 14 mg nicotine patch
  Interventions: Other: Nicotine Replacement Therapy (NRT) Sampling
- Ask, Advise, Refer (physician brief advice) (Active Comparator): Ask, Advise, Refer (physician brief advice)
  Interventions: Behavioral: Ask, Advise, Refer (physician brief advice)

INTERVENTIONS:
Other: Nicotine Replacement Therapy (NRT) Sampling — 2 week supply of 4 mg nicotine lozenge and 14 mg nicotine patch
  Arms: Nicotine Replacement Therapy (NRT)
Behavioral: Ask, Advise, Refer (physician brief advice)
  Arms: Ask, Advise, Refer (physician brief advice)

SUMMARY:
The purpose of this study is to evaluate the use of "sampling" of smoking cessation medications (nicotine patches and lozenges) among smokers seen in primary care settings. Half of study participants will be provided with samples of medication, to use however they wish; the other half will not be provided with these samples. All smokers will be advised to quit through routine contact with their physician. After the primary care contact, all participants will be contacted by phone for three brief follow-up interviews, which will involve answering questionnaires about their smoking habits.

ELIGIBILITY:
Inclusion Criteria:

* age >=18
* daily (25+ days within past 30) cigarette smoker of >5 cigs/day
* English speaking
* recruited through primary care sites aligned with study

Exclusion Criteria:

- no FDA contraindications for use of NRT:

1. not pregnant, breastfeeding, or planning to become pregnant
2. no recent (past 3 months) cardiovascular trauma: MI, stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1278 (Actual)
Dates: Start 2014-07; Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Carpenter, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Silvestri NJ, Dahne J, Wahlquist AE, Toll B, Carpenter MJ. Does Medication Sampling Improve Compliance with Brief Advice? Results from a Pragmatic Randomized Clinical Trial. J Smok Cessat. 2021;2021:6638872. doi: 10.1155/2021/6638872. Epub 2021 Mar 16. PMID 33828613

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 1,278 Enrolled:
  32 Individuals later found to be ineligible
  1 person missing contact info
  1,245 = Final Intent to Treat Sample
Groups:
- Standard Care: Ask, Advise, Refer (physician brief advice)
- Standard Care + Nicotine Replacement Therapy (NRT): 2 week supply of 4 mg nicotine lozenge and 14 mg nicotine patch + Ask, Advise, Refer (physician brief advice)
  Nicotine Replacement Therapy (NRT) Sampling: 2 week supply of 4 mg nicotine lozenge and 14 mg nicotine patch
Period: Overall Study
Arm/Group | Standard Care | Standard Care + Nicotine Replacement Therapy (NRT)
Started | 652 | 593
Completed | 652 | 593
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Standard Care + Nicotine Replacement Therapy (NRT) | Total
Number analyzed (Participants) | 652 | 593 | 1245
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (13.6) | 50.4 (13.4) | 50.7 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 365 | 391 | 756
  Male | 287 | 202 | 489
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or African American: White | 346 | 433 | 779
  White or African American: African American | 306 | 160 | 466
Heaviness of Smoking Index [Mean (Standard Deviation); unit: units on a scale] — HSI: Heaviness of Smoking Index (0-6 scale), where 6 indicates the highest ("worst") Heaviness of Smoking.
  units on a scale | 2.6 (1.6) | 2.8 (1.4) | 2.7 (1.5)
Motivation to Quit [Mean (Standard Deviation); unit: units on a scale] — Motivation to quit smoking in next month (0-10), where 0 indicates no desire to quit within the next month and 10 indicates full intent to quit within the next month.
  units on a scale | 6.2 (3.7) | 6.4 (3.6) | 6.3 (3.65)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 7-Day Self-Reported Point Prevalence Abstinence
Time Frame: From study enrollment through end of six-month follow up
Measure: Number; unit: percentage of participants
Arm/Group | Standard Care + Nicotine Replacement Therapy (NRT) | Standard Care
Number analyzed (Participants) | 593 | 652
percentage of participants | 12 | 8

2. Secondary Outcome: Any Self-defined Attempt to Stop Smoking Cigarettes
Time Frame: From study enrollment through end of six-month follow up
Measure: Number; unit: percentage of participants
Arm/Group | Standard Care + Nicotine Replacement Therapy (NRT) | Standard Care
Number analyzed (Participants) | 593 | 652
percentage of participants | 48 | 45

3. Secondary Outcome: Use of Any Smoking Cessation Medication
Time Frame: From study enrollment through end of six-month follow up
Measure: Number; unit: percentage of participants
Arm/Group | Standard Care + Nicotine Replacement Therapy (NRT) | Standard Care
Number analyzed (Participants) | 593 | 652
percentage of participants | 25 | 14

ADVERSE EVENTS:
Time Frame: Study consists of 3 follow-up phone calls at 1 month, 3 months, and 6 months post-baseline clinic visit. Adverse events are asked systematically of both groups, at all three follow-up calls.
Description: Adverse Events were monitored/assessed without regard to a specific Adverse Event Term.
Arm/Group | Standard Care | Standard Care + Nicotine Replacement Therapy (NRT)
All-Cause Mortality (participants affected / at risk) | 3/652 | 1/593
Serious Adverse Events (participants affected / at risk) | 20/652 | 9/593
Other Adverse Events (participants affected / at risk) | 289/652 | 276/593
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=652) | Standard Care + Nicotine Replacement Therapy (NRT) (N=593)
Surgical and medical procedures (Surgical and medical procedures) | 20 (22) | 9 (9)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=652) | Standard Care + Nicotine Replacement Therapy (NRT) (N=593)
Other (General disorders) | 289 (625) | 276 (596)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT02096029/Prot_SAP_000.pdf